CLINICAL TRIAL: NCT04618263
Title: A Randomized Double-blind, Placebo-controlled Single and Multiple Intravenous Ascending Dose Study of the Safety, Tolerability and Pharmacokinetics of GATE-101 in Normal Healthy Volunteers
Brief Title: Safety and Tolerability of Single and Multiple Ascending Doses of GATE-101 in Normal Human Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Reached biomarker endpoint
Sponsor: Syndeio Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GATE-101-C-101
Record Dates: First submitted 2020-10-31; First posted 2020-11-05 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Major Depressive Disorder; Excessive Sleepiness
Keywords: Major Depressive Disorder; Excessive Sleepiness; Metabotropic Glutamate Type 2/3 Receptor Antagonist
MeSH Terms: conditions — Depressive Disorder, Major; Disorders of Excessive Somnolence

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple, Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- GATE-101, 5 mg IV, Single Dose (Experimental): GATE-101, 5 mg IV, Single Dose, with follow up of 28 days
  Interventions: Drug: GATE-101
- GATE-101, 15 mg IV, Single Dose (Experimental): GATE-101, 15 mg IV, Single Dose, with follow up of 28 days
  Interventions: Drug: GATE-101
- GATE-101, 50 mg IV, Single Dose (Experimental): GATE-101, 50 mg IV, Single Dose, with follow up of 28 days
  Interventions: Drug: GATE-101
- GATE-101, 150 mg IV, Single Dose (Experimental): GATE-101, 150 mg IV, Single Dose, with follow up of 28 days
  Interventions: Drug: GATE-101
- GATE-101, 450 mg IV, Single Dose (Experimental): GATE-101, 450 mg IV, Single Dose, with follow up of 28 days
  Interventions: Drug: GATE-101
- GATE-101, 15 mg IV, Single Dose, Lumbar Catheter (Experimental): GATE-101, 15 mg IV, Single Dose, with Lumbar Catheter for collection of cerebrospinal fluid (CSF) PK samples, with follow up of 28 days
  Interventions: Drug: GATE-101
- GATE-101, 50 mg IV, Single Dose, Lumbar Catheter (Experimental): GATE-101, 50 mg IV, Single Dose, with Lumbar Catheter for collection of cerebrospinal fluid (CSF) PK samples, with follow up of 28 days
  Interventions: Drug: GATE-101
- GATE-101 5 mg IV, Five Daily Doses (Experimental): GATE-101 5 mg IV, Five Daily Doses, with follow up for 28 days from first dose
  Interventions: Drug: GATE-101
- GATE-101 15 mg IV, Five Daily Doses (Experimental): GATE-101 15 mg IV, Five Daily Doses, with follow up for 28 days from first dose
  Interventions: Drug: GATE-101
- GATE-101 150 mg IV, Five Daily Doses (Experimental): GATE-101 150 mg IV, Five Daily Doses, with follow up for 28 days from first dose
  Interventions: Drug: GATE-101
- Placebo Comparator, Single Dose (Placebo Comparator): Placebo Comparator, Single Dose, with follow up for 28 days
  Interventions: Drug: GATE-101
- Placebo Comparator, Five Daily Doses (Placebo Comparator): Placebo Comparator, Five Daily Doses, with follow up for 28 days from first dose
  Interventions: Drug: GATE-101

INTERVENTIONS:
Drug: GATE-101 — GATE-101 is a metabotropic glutamate receptor type 2/3 antagonist

SUMMARY:
To evaluate the safety, tolerability, and pharmacokinetics of single and multiple ascending doses of GATE-101 in normal human volunteers

DETAILED DESCRIPTION:
Single ascending dose (SAD), multiple ascending dose (MAD), double-blind placebo-controlled study in normal human volunteers.

Secondary objectives:

To evaluate the pharmacokinetics (PK) of GATE-101 following increasing single and multiple doses of intravenously (IV) administered GATE-101.

GATE-101 or Placebo: Dose/Mode of Administration: Single or 5 Daily Doses;Intravenous

ELIGIBILITY:
Inclusion Criteria:

1. Normal, healthy volunteer male and female subjects
2. Aged 18 to 40 years
3. For female subjects must meet one of the following:

   * Surgically sterile or at least 2 years menopausal, confirmed by follicle stimulating hormone (FSH) at screening visit, or,
   * If of childbearing potential, subject must use an acceptable method of birth control from date of screening to at least 30 days after the last dose of study drug. Must have a documented negative blood or urine pregnancy test within 24 hours prior to dosing. If reported sterile or postmenopausal, will be confirmed by FSH.
4. For male subjects, must meet one of the following:

   * Surgically sterile
   * If not surgically sterile then use of an acceptable form of contraception (condom) from the time of randomization through 30 days following the last dose of study drug. Male subjects are strongly advised to inform female partners of the need for them to use highly effective birth control during this time period.
5. Body mass index (BMI) < 30
6. Clinical laboratory values <2 times the upper limit of normal (ULN) or deemed not clinically significant by the Investigator.
7. Ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments.

Exclusion Criteria:

1. Human immunodeficiency virus (HIV) infection, or hepatitis or other ongoing infectious disease
2. Evidence of alcohol abuse (greater than 4 units of alcohol on most days; 1 unit = 1/2 pint of beer, 1 glass of wine or 1 oz. of spirits). Alcohol consumption should be avoided for at least 24 hours prior to baseline/dosing visit. A positive alcohol breathalyzer at screening and baseline visit
3. Current abuse of illicit substances, using the Diagnostic and Statistical Manual (DSM) V definition of substance use disorder.
4. Current cigarette/tobacco smoker or use of other tobacco or nicotine products including ecigarettes or vaping (if formerly a smoker must not have smoked for at least one year prior to enrolling in this study). Nonsmoking will be confirmed by cotinine assay.
5. Currently pregnant, planning to become pregnant during the course of the study, or nursing mother
6. Impaired renal function (GFR < 90 ml/min)
7. Elevated systolic blood pressure (> 130 mmHg) or diastolic blood pressure (> 80 mmHg) and/or increased QTc (>450 msec for men or >470 msec for women) or additional risk factors for Torsades de Pointes including heart failure, hypokalemia, family history of Long QT Syndrome
8. Type I or Type II diabetes
9. Malignancy in the last 5 years, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix
10. Currently taking prescription (except as listed in Section 7.4.1) or over-the-counter medications including herbal therapies, within 14 days of enrollment into the study.
11. History of allergy or sensitivity, or intolerance to NMDAR ligands including ketamine, dextromethorphan, memantine, methadone, dextropropoxyphene, or ketobemidone
12. Received another investigational drug or device within 30 days of enrollment in this study
13. Previously participated in this study
14. Psychiatric disease including major depression, bipolar disorder, anxiety, or schizophrenia, or other medical condition that, in the opinion of the Investigator, would interfere with the evaluation of study drug safety
15. For subjects in lumbar catheter Groups (6 and 7) has a history of excessive bleeding after invasive procedures or surgery or known coagulation or platelet abnormality, or has been on any blood thinner or medication affecting platelet function, such as aspirin, nonsteroidal anti-inflammatory medications, corticosteroids (except topical) or warfarin within the 7 days prior to enrollment, or has known allergy to any anesthetic agent that may be used for the lumbar puncture.
16. For subjects in lumbar catheter Groups (6 and 7) has a history of infection that required IV antibiotics within the 45 days or oral antibiotics within 30 days prior to enrollment, and, at the time of clinic admission, be febrile or have signs/symptoms consistent with an infection.
17. For subjects in lumbar catheter Groups (6 and 7) has a history of or physical examination evidence of a lumbar spine abnormality that may preclude placement of a spinal catheter, presence of intraspinal shunt devices (e.g. ventriculoperitoneal shunt), or history of elevated intracranial pressure, normal pressure hydrocephalus, or other neurological condition that in the opinion of the Investigator precludes safe study participation.
18. In the opinion of the Investigator, the Safety Monitor, or the Sponsor Study Monitor, has a history of severe renal or hepatic impairment, severe active hepatic disease, or other clinically significant medical condition that may preclude safe study participation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events Through Study Completion, 28 days | 28 Days
  Safety and Tolerabiity

SECONDARY OUTCOMES:
Pharmacokinetics - maximum plasma concentration - following a single intravenous dose | 72 hours
  Maximum observed plasma concentration following a single dose
Pharmacokinetics - maximum plasma concentration - following 5 daily intravenous doses | 72 hours
  Maximum observed plasma concentration following the fifth daily doses
Pharmacokinetics - area under the curve - following a single intravenous dose | 72 hours
  Area under the concentration time curve from time 0 to infinity following a single dose
Pharmacokinetics - area under the curve - following 5 daily intravenous doses | 72 hours
  Area under the concentration time curve from time 0 to infinity following the fifth daily dose

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Burch, MD, PhD, Study Director — Syndeio Biosciences, Inc
Locations (1):
- Clinilabs Drug Development Corporation, Eatontown, New Jersey, United States